CLINICAL TRIAL: NCT07237841
Title: Preoperative Carbohydrate Loading in Patients With Well-controlled Type 2 Diabetes Mellitus
Brief Title: Preoperative Carbohydrate Loading in Diabetes Mellitus
Acronym: PRECARB-DMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50/NDGĐ-HĐĐĐ
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Type2diabetes; Enhanced Recovery After Surgery (ERAS); Fasting; Carbohydrate Loading; Gastric Emptying
Keywords: Carbohydrate loading; Preoperative care; Gastric residual; Fasting; ERAS
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: interventional group and controlled group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard fasting group (No Intervention): Participants fast for at least six hours before anesthesia, following standard preoperative fasting guidelines.
  Capillary blood glucose is measured at baseline, and at 1, 2, and 4 hours before surgery.
- Carbohydrate loading group (25% carbohydrate solution) (Experimental): Participants receive 200 mL of 25% carbohydrate solution two hours before anesthesia.
  Capillary blood glucose is measured at baseline, and at 1, 2, and 4 hours after ingestion.
  Preoperative gastric ultrasonography is performed 2 hours after ingestion to assess residual gastric volume.
  Interventions: Dietary Supplement: 25% Carbohydrate solution (CHO drinking)

INTERVENTIONS:
Dietary Supplement: 25% Carbohydrate solution (CHO drinking) — Participants in the experimental arm will receive 200 mL of 25% carbohydrate solution (containing oligosaccharides) 2 hours before induction of anesthesia. The solution is consumed orally within 30 minutes.
  Capillary blood glucose is measured using an ACCU-CHEK Active glucometer at baseline (before ingestion), and at 1 hour, 2 hours, and 4 hours after ingestion.
  Preoperative gastric ultrasonography is performed 2 hours after ingestion in the right lateral decubitus position to estimate gastric volume and detect residual gastric content.
  If blood glucose remains > 10 mmol/L for more than 180 minutes, patients will receive intravenous insulin infusion according to the hospital's protocol.
  The purpose of this intervention is to evaluate the safety and metabolic impact of preoperative carbohydrate loading in well-controlled type 2 diabetes mellitus patients.
  Arms: Carbohydrate loading group (25% carbohydrate solution)

SUMMARY:
This prospective, randomized, open-label, parallel-group clinical trial aims to evaluate the safety and metabolic effects of preoperative carbohydrate loading in patients with well-controlled type 2 diabetes mellitus (T2DM) undergoing elective surgery.

The study is conducted at Nhan Dan Gia Dinh Hospital (Ho Chi Minh City, Vietnam) over a 20-month period (March 2023-October 2025). Eligible participants are adults aged 18-65 years with well-controlled T2DM (HbA1c <7%, fasting plasma glucose 6.5-10 mmol/L) and no risk factors for aspiration or gastroparesis.

Participants are randomly assigned to two groups: the intervention group receives 200 mL of 25% carbohydrate solution 2 hours before anesthesia, while the control group follows standard preoperative fasting. Capillary blood glucose is measured at baseline and at 1, 2, and 4 hours after ingestion. Preoperative gastric volume is assessed by bedside ultrasonography to detect residual gastric contents.

The primary outcome is capillary blood glucose level at 4 hours after carbohydrate ingestion. Secondary outcomes include total intravenous insulin used for hyperglycemia management and the proportion of patients with gastric residual volume >1.5 mL/kg.

This study hypothesizes that preoperative carbohydrate loading in well-controlled T2DM patients increases blood glucose by no more than 2 mmol/L at 4 hours after ingestion compared to fasting, without increasing gastric residual volume or aspiration risk.

The results are expected to provide additional evidence on the safety of preoperative carbohydrate loading in diabetic patients, supporting its inclusion in Enhanced Recovery After Surgery (ERAS) protocols for optimized perioperative care.

DETAILED DESCRIPTION:
Preoperative carbohydrate loading has been widely recognized as a core component of Enhanced Recovery After Surgery (ERAS) protocols. In non-diabetic patients, drinking a carbohydrate solution two hours before anesthesia improves perioperative metabolic status, reduces insulin resistance, and enhances postoperative recovery without increasing the risk of aspiration or other complications. However, its safety and effectiveness in patients with type 2 diabetes mellitus (T2DM) remain controversial due to concerns about delayed gastric emptying and hyperglycemia.

Recent studies have shown that preoperative carbohydrate drinks in patients with well-controlled T2DM do not significantly delay gastric emptying and cause only transient increases in blood glucose levels, typically returning to baseline within 180 minutes. These findings suggest that carbohydrate loading may be safe for this population, provided their diabetes is well managed and they have no symptoms of gastroparesis. Despite this, current guidelines remain cautious, and further evidence is needed to strengthen clinical recommendations, particularly in Asian populations.

This randomized, open-label, parallel-group clinical trial is being conducted at Nhan Dan Gia Dinh Hospital, Ho Chi Minh City, Vietnam. The study enrolls adult patients (aged 18-65 years) with well-controlled T2DM (HbA1c <7%, fasting glucose 6.5-10 mmol/L) scheduled for elective surgery under general anesthesia. Participants are randomly assigned in a 1:1 ratio to receive either 200 mL of 25% carbohydrate solution two hours before anesthesia (intervention group) or to continue standard fasting for at least six hours before surgery (control group). Randomization is performed using computer-generated allocation.

Capillary blood glucose levels are measured at baseline and at 1, 2, and 4 hours after ingestion. Bedside gastric ultrasonography is used to estimate gastric volume before anesthesia, and residual volume greater than 1.5 mL/kg is considered gastric retention. Patients with capillary glucose >10 mmol/L persisting beyond 180 minutes will receive intravenous insulin infusion according to the hospital protocol.

The primary endpoint is capillary blood glucose level at four hours after carbohydrate ingestion. Secondary outcomes include total insulin administered to treat hyperglycemia and the proportion of participants with gastric retention before anesthesia. Safety outcomes include incidence of aspiration, diabetic ketoacidosis, and other adverse events.

The hypothesis is that preoperative carbohydrate loading in well-controlled T2DM increases blood glucose by no more than 2 mmol/L compared with fasting and does not increase gastric residual volume or aspiration risk. If confirmed, these findings will provide new evidence supporting the safe integration of carbohydrate loading into ERAS protocols for diabetic patients, helping to improve comfort, reduce perioperative stress, and optimize recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years scheduled for elective surgery under general anesthesia.
* Diagnosed with type 2 diabetes mellitus with well-controlled glycemia (HbA1c < 7% within the last 3 months).
* Fasting plasma glucose between 6.5 and 10 mmol/L on the day before surgery.
* ASA physical status II-III.
* Capable of oral intake and able to provide written informed consent.
* No contraindication to carbohydrate ingestion or ultrasonographic gastric assessment.

Exclusion Criteria:

* History or clinical evidence of gastroparesis, gastroesophageal reflux disease (GERD), or hiatal hernia.
* Conditions increasing aspiration risk: obesity (BMI > 30 kg/m²), pregnancy, or emergency surgery.
* Severe systemic comorbidities (renal failure, hepatic failure, heart failure, or COPD exacerbation).
* Use of medications affecting gastric motility (opioids, prokinetics, anticholinergics) within 24 hours.
* Known hypersensitivity or intolerance to carbohydrate drink components.
* Refusal or inability to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose level (mmol/L) at 4 hours after carbohydrate ingestion | 4 hours post-ingestion
  Measured by capillary blood sample using ACCU-CHEK Active device. The endpoint tests the non-inferiority hypothesis that glucose elevation does not exceed +2 mmol/L compared to the control group.

SECONDARY OUTCOMES:
Capillary blood glucose levels at 1 and 2 hours after ingestion | 1 and 2 hours post ingestion
Total intravenous insulin administered for hyperglycemia (>10 mmol/L) | Up to 4 hours after ingestion
Proportion of patients with gastric retention (GV/W >1.5 mL/kg) | Preoperative (2 hours after ingestion)

CONTACTS AND LOCATIONS:
Overall Officials: Huynh Van Binh, Study Director — Nhan dan Gia Dinh Hospital
Locations (1):
- Binh Huynh, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustafsson UO, Nygren J, Thorell A, Soop M, Hellstrom PM, Ljungqvist O, Hagstrom-Toft E. Pre-operative carbohydrate loading may be used in type 2 diabetes patients. Acta Anaesthesiol Scand. 2008 Aug;52(7):946-51. doi: 10.1111/j.1399-6576.2008.01599.x. Epub 2008 Mar 7. PMID 18331374